CLINICAL TRIAL: NCT05789108
Title: Deep Venous Thrombosis and Risk of Long Term Complications in Acutely Admitted Patients
Brief Title: Deep Venous Thrombosis and Long Term Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ove Andersen (Other)
Responsible Party: Sponsor-Investigator, Ove Andersen, Research Director and Head of the Department of Clinical Research, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-21061004 / 85280
Record Dates: First submitted 2023-02-13; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: DVT of Legs
Keywords: DVT; aging; inflammation; anti-inflammation; immune system; PTS
MeSH Terms: conditions — Venous Thrombosis; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biomarkers and long term complications in DVT patients (Other): Patients with DVT will be enrolled in the study during their hospitalization at the ED. The enrolled patients will have 4 follow-up visits, 1) during the first 14 days after diagnosis, 2) after 3 months, 3) after 12 months and 4) 24 months after the time of diagnosis.
  Interventions: Diagnostic Test: Blood sample and Ultrasound examination

INTERVENTIONS:
Diagnostic Test: Blood sample and Ultrasound examination — The ultrasound examination is a non-invasive procedure with no risks, adverse reactions, or discomforts associated with the examination. The study blood samples are mostly obtained at the same time as clinical blood sample collection in order to avoid unnecessary complications.
  The inclusion and ultrasound examiniation is performed by the patient responsible physician at the Emergency Department. Blood samples during the study period are performed by trained study staff.

SUMMARY:
In this cohort study, the investigators will investigate the concentration of biomarkers, e.g., inflammatory, anti-inflammatory, immunological, senescent, biochemical ratio-calculations and blood cell type among first time lower extremity deep venous thrombosis patients with and without SARS-CoV-2 infection and long term complications with a 2-year follow-up.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) which is a common concept for deep venous thrombosis (DVT) and pulmonary embolus (PE) is the third most common cardiovascular disease after myocardial infarction and stroke. The incidence of deep venous thrombosis (DVT) increases exponentially with age and is highest in high-income countries compared to low-income countries. The pathophysiology of DVT is of multicomplex aetiology and there are multifactorial causes leading to the development of DVT. In the long term, patients with DVT can experience reduced thrombus resolution, recurrent thrombosis, and post thrombotic syndrome (PTS), where inflammation has a major impact.

The investigators hypothesis are:

i. There is an increased level of biomarkers at time of diagnosis among DVT patients who develop PTS compared to DVT patients who do not develop PTS

ii. There is an elevated level of the biomarkers: suPAR, D-dimer, inflammatory, anti-inflammatory, immunological, and aging markers at the time of diagnosis of DVT in patients with SARS-CoV-2 infection compared to DVT patients without SARS-CoV-2 infection.

iii. There is an increased incidence of late complications such as PTS among DVT patients with SARS-CoV-2 infection compared to DVT patients without SARS-CoV-2 infection

Purpose:

In this clinical prospective cohort study the investigators will investigate and characterize acutely admitted patients with deep venous thrombosis via inflammatory, anti-inflammatory, immunological and ageing biomarkers to gain a better understanding of options about prevention and treatment of long-term complications

Data collection:

Eligible patients will be included in the Emergency Department by the physician responsible for the treatment.

Variables:

The following variables will be collected at inclusion and 4 follow-up visits: information on demographics, biomarkers (blood samples and ultrasound scan), clinical data from the patient case report, self-reported information on risk factors, socioeconomic variables, quality of life, and pain. Moreover, register data on socioeconomic status, morbidity, physical health by e.g. Charlson score, mortality, hospital visits, and prescriptions will be retrieved after 2 years of follow-up.

Sample size:

To detect a difference in suPAR (0-24 months) and the association between suPAR and the risk of developing PTS (0-24 months) a total of 150 participants are needed in the study.

The collected data will be kept in accordance with the Data Protection Agency guidelines. The studies are carried out in accordance with the principles of the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above
* First time lower extremity DVT
* Hospitalized at the Emergency Department

Exclusion Criteria:

* Patients without a Danish social security number
* Terminal patients
* Patients who do not understand or speak Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
suPAR - baseline | Baseline
  suPAR level in first-time DVT patients at the time of diagnosis (baseline)
Change in suPAR - 90 days | 90 days
  Change in suPAR level in first-time DVT patients from the time of diagnosis (baseline) to 90 days
Change in suPAR - 12 months | 12 months
  Change in suPAR level in first-time DVT patients from the time of diagnosis (baseline) to 12 months
Change in suPAR - 24 months | 24 months
  Change in suPAR level in first-time DVT patients from the time of diagnosis (baseline) to 24 months
Association of suPAR and PTS - baseline | Baseline
  Association of suPAR and development of PTS in DVT patients from the time of diagnosis (baseline)
Association of suPAR and PTS - 90 days | 90 days
  Association of suPAR and development of PTS in DVT patients from the time of diagnosis and 90 days after diagnosis
Association of suPAR and PTS - 12 month | 12 months
  Association of suPAR and development of PTS in DVT patients from the time of diagnosis and 12 months after diagnosis
Association of suPAR and PTS - 24 month | 24 months
  Association of suPAR and development of PTS in DVT patients from the time of diagnosis and 24months after diagnosis

SECONDARY OUTCOMES:
Biomarkers in DVT patients - baseline | Baseline
  Biomarkers concerning inflammatory, anti-inflammatory, immunological and aging/ senescent cells (IL-1β, IL-6, IL-10, IL-15, IL-18, Trombin, Fibrin/ Fibrinogen, GDF-8, GDF-15, COX2, PGE2, CD57, Cystatin C, NGAL, FGF-21, FGF-23, MICA, ULBP2, Klotho, p16INK4a, p21Cip1, asparagine endopeptidase, DPP4, KLRG1, DNA-methylering, U-PA, Vitronectin, PAI-1, Tissue Factor, histoner, kromatin and NETs) at baseline.
Biomarkers in DVT patients - change over time 90 days | 90 days
  Change in biomarkers concerning inflammatory, anti-inflammatory, immunological and aging/ senescent cells (IL-1β, IL-6, IL-10, IL-15, IL-18, Trombin, Fibrin/ Fibrinogen, GDF-8, GDF-15, COX2, PGE2, CD57, Cystatin C, NGAL, FGF-21, FGF-23, MICA, ULBP2, Klotho, p16INK4a, p21Cip1, asparagine endopeptidase, DPP4, KLRG1, DNA-methylering, U-PA, Vitronectin, PAI-1, Tissue Factor, histoner, kromatin and NETs) from time of diagnosis (baseline) to 90 days after diagnosis.
Biomarkers in DVT patients - change over time 12 months | 12 months
  Change in biomarkers concerning inflammatory, anti-inflammatory, immunological and aging/ senescent cells (IL-1β, IL-6, IL-10, IL-15, IL-18, Trombin, Fibrin/ Fibrinogen, GDF-8, GDF-15, COX2, PGE2, CD57, Cystatin C, NGAL, FGF-21, FGF-23, MICA, ULBP2, Klotho, p16INK4a, p21Cip1, asparagine endopeptidase, DPP4, KLRG1, DNA-methylering, U-PA, Vitronectin, PAI-1, Tissue Factor, histoner, kromatin and NETs) from time of diagnosis (baseline) to 12 months after diagnosis.
Biomarkers in DVT patients - change over time 24 months | 24 months
  Change in biomarkers concerning inflammatory, anti-inflammatory, immunological and aging/ senescent cells (IL-1β, IL-6, IL-10, IL-15, IL-18, Trombin, Fibrin/ Fibrinogen, GDF-8, GDF-15, COX2, PGE2, CD57, Cystatin C, NGAL, FGF-21, FGF-23, MICA, ULBP2, Klotho, p16INK4a, p21Cip1, asparagine endopeptidase, DPP4, KLRG1, DNA-methylering, U-PA, Vitronectin, PAI-1, Tissue Factor, histoner, kromatin and NETs) from time of diagnosis (baseline) to 24 months after diagnosis.
PTS in DVT patients - 90 days | 90 days
  Development of PTS in DVT patients from the time of diagnosis (baseline) and up to 90 days after diagnosis.
PTS in DVT patients - 12 months | 12 months
  Development of PTS in DVT patients from the time of diagnosis (baseline) and up to 12 months after diagnosis.
PTS in DVT patients - 24 months | 24 months
  Development of PTS in DVT patients from the time of diagnosis (baseline) and up to 24 months after diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, M.D., Ph.D., Principal Investigator — Department of Clinical Research; Izzet Altintas, M.D., Study Chair — Department of Clinical Research
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No